CLINICAL TRIAL: NCT05028413
Title: Pilot Randomized Control Trial of Smartphone-enabled Breath Alcohol Monitoring on Perceived Fitness to Drive a Vehicle Among Intoxicated Adults
Brief Title: Evaluating Perceived Fitness to Drive While Intoxicated
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, M. Kit Delgado, MD, Assistant Professor of Emergency Medicine and Epidemiology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 827284
Record Dates: First submitted 2021-08-24; First posted 2021-08-31 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Drinking; Alcohol Intoxication; Perception, Self; Drinking, Alcohol; Driving Under the Influence; Drinking Behavior
MeSH Terms: conditions — Alcohol Drinking; Alcoholic Intoxication; Driving Under the Influence; Drinking Behavior | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants Blinded to BrAC reading (Control) (No Intervention): Participants randomized to this arm will consume three weight-based doses of alcohol with a target BAC of 0.10 and comple breathalyzer measurements every 20 minutes until a BAC of 0.03 is reached. They will complete a visual analog scale (the Self-Reported intoxication Survey) on their perceived fitness to drive and be blinded to their breath alcohol readings with the BACtrack Mobile Pro device.
- Participants Aware of their BrAC reading (Experimental): Participants randomized to this arm will consume three weight-based doses of alcohol with a target BAC of 0.10 and comple breathalyzer measurements every 20 minutes until a BAC of 0.03 is reached. They will be shown their breath alcohol readings with the BACtrack Mobile Pro device before completing a visual analog scale (the Self-Reported intoxication Survey) on their perceived fitness to drive.
  Interventions: Behavioral: Participants Shown their Breath Alcohol Content Measurement

INTERVENTIONS:
Behavioral: Participants Shown their Breath Alcohol Content Measurement — Each time a Breath Alcohol Content (BrAC) Measurement is taken by the research team, the participant is shown the measurement before completing the paper visual analog scale scale (the Self-Reported intoxication Survey) on their perceived fitness to drive.
  Arms: Participants Aware of their BrAC reading

SUMMARY:
The goal of this study is to conduct a laboratory-based pilot randomized control trial of smartphone-enabled breath alcohol monitoring on perceived fitness to drive a vehicle among intoxicated adults. The study team will enroll up to 30 adults aged > 21-44 who are frequent drinkers without dependence who drive more than four times per week to complete a standardized alcohol drinking protocol in a monitored setting collecting breathalyzer measurements. The protocol involves consuming three weight-based doses of alcohol with a target BAC of 0.10 and completing breathalyzer measurements every 20 minutes until a BAC of 0.03 is reached. The control group will complete a visual analog scale on their perceived fitness to drive and be blinded to their breath alcohol readings with the BACtrack Mobile Pro breathalyzer device, while the intervention group would do the same, but be shown their breath alcohol readings on the paired BACtrack smartphone application. The research team's previous research has validated the accuracy of the BACtrack Mobile Pro device to measure BAC within +/- 0.001 of police-grade breathalyzer and estimate BAC within +/- 0.01 of a blood test.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-39 years old,
* Less than 4 drinking days and less than 12 drinks per week on average in the past 2 months,
* Have consumed at least 4 (women) or 5 (men) drinks on one occasion, in the past year without experiencing adverse effects
* Have a valid photo ID
* Willing and able to use a rideshare credit or septa token as transportation home from the study visit
* Drives at least 2 days per week on average.

Exclusion Criteria:

* Desire alcohol treatment now or received it in the past 6 months,
* Have Alcohol use disorder per DSM-V criteria
* Meet or have met criteria for a substance use disorder within the past 12 months per DSM V criteria
* Have a prior psychiatric condition requiring hospitalization
* Are non-English-speaking
* Individuals who have a medical condition or who are taking medication which limits or prevents the consumption of alcohol
* Are experiencing suicidal ideation

Ages: 21 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harrison EL, Marczinski CA, Fillmore MT. Driver training conditions affect sensitivity to the impairing effects of alcohol on a simulated driving test [corrected]. Exp Clin Psychopharmacol. 2007 Dec;15(6):588-98. doi: 10.1037/1064-1297.15.6.588. PMID 18179312
- [Background] Harrison EL, Fillmore MT. Are bad drivers more impaired by alcohol? Sober driving precision predicts impairment from alcohol in a simulated driving task. Accid Anal Prev. 2005 Sep;37(5):882-9. doi: 10.1016/j.aap.2005.04.005. PMID 15907777
- [Background] Marczinski CA, Stamates AL. Artificial sweeteners versus regular mixers increase breath alcohol concentrations in male and female social drinkers. Alcohol Clin Exp Res. 2013 Apr;37(4):696-702. doi: 10.1111/acer.12039. Epub 2012 Dec 6. PMID 23216417
- [Background] McCarthy DM, Niculete ME, Treloar HR, Morris DH, Bartholow BD. Acute alcohol effects on impulsivity: associations with drinking and driving behavior. Addiction. 2012 Dec;107(12):2109-14. doi: 10.1111/j.1360-0443.2012.03974.x. Epub 2012 Aug 10. PMID 22690907
- [Background] Patton JH, Stanford MS, Barratt ES. Factor structure of the Barratt impulsiveness scale. J Clin Psychol. 1995 Nov;51(6):768-74. doi: 10.1002/1097-4679(199511)51:63.0.co;2-1. PMID 8778124
- [Background] Senecal N, Wang T, Thompson E, Kable JW. Normative arguments from experts and peers reduce delay discounting. Judgm Decis Mak. 2012 Sep 1;7(5):568-589. PMID 23596504
- [Derived] Ebert JP, Kranzler HR, Barnett IJ, Hemmons JE, Yan R, Spencer E, Delgado MK. Effect of smartphone breathalyzer feedback on willingness to drive in moderately intoxicated individuals: A randomized trial. Psychol Addict Behav. 2025 Nov;39(7):669-675. doi: 10.1037/adb0001088. Epub 2025 Aug 14. PMID 40811123
- See also: BacTrack Mobile Smartphone Paired Breathalyzer — https://www.bactrack.com/products/bactrack-mobile-smartphone-breathalyzer

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants Blinded to BrAC Reading (Control) | Participants Aware of Their BrAC Reading
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 20 patients analyzed between the ages of 21 and 39 that have a driver's license and have consumed alcohol (4 or more drinks for a woman)/ ( or more drinks or men) in on driving occasion without any problems. Participants have not received alcohol treatment in the last 6 months, do not desire alcohol treatment, nor are pregnant or nursing.
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Blinded to BrAC Reading (Control) | Participants Aware of Their BrAC Reading | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.7 (4.2) | 28.5 (4.2) | 27.1 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: White | 7 | 9 | 16
  United States: Asian | 3 | 0 | 3
  United States: Black | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Participants' Perceived Fitness to Drive Measurement
Description: Participant's self rating on visual analog scale from 1-10 (1: Extremely Able to Drive; 10: Not at all Able to Drive) after Breath Alcohol Content Measurement was collected
Time Frame: The duration of study visit, up to 8 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Blinded to BrAC Reading (Control) | Participants Aware of Their BrAC Reading
Number analyzed (Participants) | 10 | 10
units on a scale | 6.5 (2.5) | 4.6 (1.9)

2. Secondary Outcome: Participants' Perceived Willingness to Drive Measurement
Description: Participant's self rating on visual analog scale from 1-10 (1: Not at all Willing to Drive; 10: Extremely Willing to Drive) after Breath Alcohol Content Measurement was collected
Time Frame: The duration of study visit, up to 8 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Blinded to BrAC Reading (Control) | Participants Aware of Their BrAC Reading
Number analyzed (Participants) | 10 | 10
units on a scale | 3.5 (2.3) | 5.5 (2.5)

ADVERSE EVENTS:
Time Frame: 8 hours
Description: Screening for eligibility reduced risk of all risk mortality
Arm/Group | Participants Blinded to BrAC Reading (Control) | Participants Aware of Their BrAC Reading
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT05028413/Prot_SAP_000.pdf